CLINICAL TRIAL: NCT02315404
Title: Cap Assisted Balloon Enteroscopy Versus Conventional Balloon Enteroscopy In The Evaluation Of Obscure Gastrointestinal Bleeding: A Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor Enrollment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SBE CAP 1
Record Dates: First submitted 2014-01-06; First posted 2014-12-11 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Obscure Gastrointestinal Bleeding
Keywords: Obscure gastrointestinal bleeding; Overt gastrointestinal bleeding; Occult gastrointestinal bleeding; Enteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No cap (Placebo Comparator): enteroscopy performed without a cap
  Interventions: Procedure: CAP
- Enteroscopy with a cap (Active Comparator): Enteroscopy performed with a CAP fitted to the end of the scope
  Interventions: Procedure: CAP

INTERVENTIONS:
Procedure: CAP — CAP fitted to the end of the endoscope

SUMMARY:
Gastrointestinal bleeding originating from the small bowel is difficult to diagnose and treat because the small bowel is difficult to see and reach. Balloon assisted enteroscopy (BAE) is a new enteroscopy methods that allow examination of the small bowel and allows for diagnosis and treatment of bleeding originating from this part of the intestine. Unfortunately, BAE is unsuccessful in identifying the cause of bleeding in 40-50% of patients. This may be due to limited visualization of the small bowel lining during conventional endoscopy. One way to improve visualization of the small bowel lining is by adding a transparent plastic cap to the end of the endoscope (camera), which allows the endoscope to see around sharp turned and behind folds in the small bowel.

The investigators goal in this randomized controlled study is to see if adding a transparent cap to the end of the endoscope will help to identify and treat small bowel bleeding. The investigators will invite patients referred for BAE to participate in the study; the alternative to participating in the study is having standard BAE (without a cap). If patients choose to participate in the study they will be randomized to BAE with or without a cap on the end of the endoscope. Subjects time commitment will be limited to the consent process and pre-procedure paperwork at time of initial endoscopy and time required to complete telephone questionnaire at 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old) patients undergoing BAE for the evaluation of OGIB or iron deficiency anemia.

Exclusion Criteria:

* Unable to provide written informed consent.
* Pregnancy or lactation.
* Suspected bowel obstruction or GI perforation.
* Unable to tolerate sedation or general anesthesia due to medical co-morbidities.
* Uncorrected coagulopathy (platelet count <50,000, INR> 2, PTT> 2x upper limit of normal).
* Patient undergoing retrograde BAE.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-01; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of BAE vs. Cap assisted BAE (C-BAE). | 1 day
  Diagnostic yield defined as proportion of enteroscopies in which clinically significant findings were identified.
  a. Clinically significant findings being defined as P2 lesion (lesion considered to have high potential for bleeding; such as typical angiomata, large ulceration, tumor or varices)

SECONDARY OUTCOMES:
Overall Diagnostic yield of BAE vs. C-BAE | 1 day
  Diagnostic yield defined as proportion of enteroscopies in which any abnormality is detected.
  a. Abnormalities classified as: i. P0: lesion with no bleeding potential, including visible submucosal veins, diverticula without the presence of blood or nodules without mucosal break.
  ii. P1: lesion considered as having uncertain bleeding potential, such as a red spot on the intestinal mucosa or small erosions.
  iii. P2: lesion considered to have high potential for bleeding; such as typical angiomata, large ulceration, tumor or varices
Therapeutic yield BAE vs. Cap assisted BAE (C-BAE). | 1 day
  Therapeutic yield being defined as proportion of enteroscopies in which a therapeutic intervention was undertaken. Interventions included in this calculation were polypectomy, argon plasma coagulation, bipolar coagulation, dilation of strictures, and endoscopic clipping. Biopsy was considered to be a therapeutic intervention if histopathology results lead to the initiation of a medical or surgical therapy (i.e: resection of mass, medical therapy for Crohn's disease)
iii. Depth of small bowel insertion: calculated according to the method of Efthymiou et al. | 1 day
  Fold counting method: The number of complete folds (valvulae conniventes) will be counted during withdrawal of the endoscope; with the assumption that the distance between folds is approximately 0.9 cm.
vProcedure related adverse events. | 1 day
Recurrence of GI bleeding at 12 months, as evaluated by questionnaire | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States